CLINICAL TRIAL: NCT00067015
Title: Phase III Randomized Trial Study Comparing the Outcome of High-Dose IMRT (86.4 GY) Alone With IMRT to 75.6 GY Plus Neoadjuvant/Adjuvant Androgen Deprivation in Patients With High Grade Intermediate Risk and Unfavorable Risk Prostate Cancer
Brief Title: Radiation Therapy With or Without Bicalutamide and Goserelin in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03-040; P30CA008748 (NIH); MSKCC-03040
Record Dates: First submitted 2003-08-08; First posted 2003-08-11 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide; Goserelin; Radiotherapy

ARMS (2):
- IMRT alone to 86.4 Gy (Experimental): External radiotherapy is given for 10 weeks, Monday through Friday for a total of 48 sessions. The total dose of radiotherapy delivered during these 10 weeks is 86.4 Gy. The radiation treatments are delivered with a high precision technique called intensity modulated radiotherapy or IMRT. For this treatment, no hormonal therapy is required.
  Interventions: Procedure: assessment of therapy complications; Procedure: quality-of-life assessment; Radiation: radiation therapy
- IMRT TO 75.6 Gy plus Adjuvant Androgen Deprivation (Experimental): Prior to a planned course of radiotherapy, which will last for eight and a half weeks, 10 weeks of hormonal therapy are given. The hormonal therapy will start with a daily pill called Casodex. Three to seven days after starting this pill, a Zoladex injection will be administered in addition to the Casodex pill. Zoladex hormonal therapy is given in the form of a monthly injection. After 10 weeks from the initiation of hormone therapy, you will begin external radiotherapy. For these treatments only 42 treatment sessions are given. The total dose of radiotherapy delivered during these 8.5 weeks is 75.6 Gy. The hormone injections continue during the radiation treatments and for 2 years after the radiation treatments. The pills are only taken for the 10 weeks before and also during the radiation treatments, however afterwards the pills are discontinued.
  Interventions: Drug: bicalutamide; Drug: goserelin acetate; Procedure: assessment of therapy complications; Procedure: quality-of-life assessment; Radiation: radiation therapy

INTERVENTIONS:
Drug: bicalutamide
  Arms: IMRT TO 75.6 Gy plus Adjuvant Androgen Deprivation
Drug: goserelin acetate
  Arms: IMRT TO 75.6 Gy plus Adjuvant Androgen Deprivation
Procedure: assessment of therapy complications
Procedure: quality-of-life assessment
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Giving radiation therapy in different ways may cause less damage to normal tissue and may improve quality of life and help patients live more comfortably. Androgens can stimulate the growth of prostate cancer cells. Drugs such as goserelin and bicalutamide may fight cancer by stopping the production of androgens. It is not yet known whether radiation therapy is more effective with or without goserelin and bicalutamide in treating prostate cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of high-dose radiation therapy with or without bicalutamide and goserelin in treating patients who have prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the quality of life of patients with high-grade intermediate-risk or unfavorable-risk adenocarcinoma of the prostate when treated with high-dose intensity-modulated radiotherapy alone versus with androgen deprivation comprising bicalutamide and goserelin.
* Compare the prostate-specific antigen relapse-free, distant metastases-free, and overall survival of patients treated with these regimens.
* Compare the toxicity of these regimens in these patients.
* Compare the local control in patients treated with these regimens, based on post-treatment sextant biopsies performed 4 years after study completion.

OUTLINE: This is a randomized study. Patients are stratified according to prostate-specific antigen level, Gleason score, and clinical stage. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo high-dose intensity-modulated radiotherapy (IMRT) 4-5 times per week for 10 weeks (a total of 48 treatments).
* Arm II: Patients receive oral bicalutamide once daily for 18.5 weeks. Three to seven days after the initiation of bicalutamide, patients also receive goserelin subcutaneously monthly for 2 years. Beginning after 10 weeks of hormonal therapy, patients undergo concurrent high-dose IMRT 4-5 times per week for 8.5 weeks (a total of 42 treatments). Patients discontinue bicalutamide on or near the end of radiotherapy.

In both arms, treatment continues in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, every 3 months for 1.5 years after the completion of radiotherapy, then 6 months later, and then annually for 2 years.

Patients are followed every 6-8 months for 4 years and then annually for 2 years.

PROJECTED ACCRUAL: A total of 400 patients (200 per treatment arm) will be accrued for this study within 4-5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate
* Unfavorable-risk disease, including at least 2 of the following characteristics:

  * Prostate-specific antigen level greater than 10 ng/mL
  * Gleason score greater than 7
  * Stage T4
* Intermediate-risk disease with a Gleason score of at least 8 allowed
* Lymph nodes clinically negative by imaging studies or histologically negative by node sampling or lymph node dissection
* Prostate size less than 75 grams
* No distant metastases by bone scan, CT scan, or MRI

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 80-100%

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT and SGPT no greater than 1.5 times ULN

Renal

* Not specified

Other

* No documented history of inflammatory bowel disease
* No bilateral hip replacements
* No other invasive cancer except localized basal cell or squamous cell skin cancer unless disease free for at least 5 years
* No major medical or psychiatric illness that would preclude study completion, compliance, or follow-up

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy for prostate cancer

Endocrine therapy

* No prior androgen-deprivation therapy

Radiotherapy

* No prior pelvic radiotherapy
* No prior prostate brachytherapy

Surgery

* No prior bilateral orchiectomy
* No prior radical prostatectomy
* No prior cryotherapy for prostate cancer

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2003-05; Primary Completion 2004-10 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
compare the quality of life | 2 years

SECONDARY OUTCOMES:
response | 2 years
toxicity | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Zelefsky, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States